CLINICAL TRIAL: NCT05799495
Title: A PHASE 2B, DOUBLE-BLIND, RANDOMIZED, PLACEBO-CONTROLLED, PARALLEL GROUP, DOSE RANGING STUDY TO EVALUATE VIROLOGICAL RESPONSE AND SAFETY OF ORAL PF-07817883 IN NON-HOSPITALIZED SYMPTOMATIC ADULT PARTICIPANTS WITH COVID-19
Brief Title: A Study to Understand the Effect and Safety of the Study Medicine PF-07817883 in Adults Who Have Symptoms of COVID-19 But Are Not Hospitalized
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C5091003; 2022-002871-12 (EudraCT Number); 2023-506667-34-00 (EU CTIS Number)
Record Dates: First submitted 2023-04-04; First posted 2023-04-05 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-09

CONDITIONS: SARS-CoV-2 Infection
Keywords: COVID-19; SARS COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1: low dose (Experimental)
  Interventions: Drug: PF-07817883
- Arm 2: medium dose (Experimental)
  Interventions: Drug: PF-07817883
- Arm 3: high dose (Experimental)
  Interventions: Drug: PF-07817883
- Arm 4: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-07817883 — Arm 1: low dose Arm 2: medium dose Arm 3: high dose
  Arms: Arm 1: low dose; Arm 2: medium dose; Arm 3: high dose
Drug: Placebo — Placebo
  Arms: Arm 4: Placebo

SUMMARY:
The purpose of the study is to understand the effects and safety of PF-07817883 treatment. The study wants to know how PF-07817883 treatment lowers the level of the virus that causes COVID 19. To understand that samples are collected from adult participants who have the symptoms of COVID 19 but are not hospitalized.

The study is seeking for participants who:

* are 18 years of age or older at the time of entering the study.
* have a positive rapid antigen test within 48 hours before entering the study. Rapid antigen test is a test done to confirm the presence of a specific virus in the body.
* have onset of signs or symptoms of COVID-19 within 5 days before entering the study.
* have at least 1 of the specified signs or symptoms of COVID-19 present on the day of entering the study.

Around 228 participants with a confirmed case of COVID 19 are planned to be taken into the study. Participants will be randomly grouped to receive PF-07817883. Three groups will receive 100, 300, 600mg of PF-07817883 and one of the groups will receive placebo (a pill that doesn't have any medicines) orally every 12 hours for 5 days.

The study is going to last up to 5 weeks. This includes the initial period of selecting participants, participants receiving the medicine or the placebo and then a 4-week follow-up period after giving the participants the last medicine.

The study team will monitor how each participant is doing with the study treatment during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Participants ≥18 to <65 years of age at the time of the Screening Visit.

   * WOCBP may be enrolled.
   * All fertile participants must agree to use a highly effective method of contraception.
2. Confirmed SARS-CoV-2 infection as determined by RAT in NP specimen collected within 48 hours prior to randomization. Investigator sites will use test kits that are authorized for use in this study and the test result must be available to confirm eligibility.
3. Initial onset of signs/symptoms attributable to COVID-19 within 5 days prior to the day of randomization and at least 1 of the specified signs/symptoms attributable to COVID-19 present on the day of randomization.

Exclusion Criteria:

1. Current need for hospitalization or anticipated need for hospitalization within 24h after randomization in the clinical opinion of the site investigator.
2. Known medical history of active liver disease (other than nonalcoholic hepatic steatosis), including chronic or active hepatitis B or C infection, primary biliary cirrhosis, Child-Pugh Class B or Class C, or acute liver failure.
3. History of hypersensitivity or other contraindication to any of the components of the study interventions, as determined by the investigator.
4. Suspected or confirmed concurrent active systemic infection other than COVID-19 that may interfere with the evaluation of response to the study intervention.
5. Immunocompromised with ≥1 of the following:

   1. Solid organ (eg, liver, heart, lung or kidney) transplant recipient who is receiving immunosuppressive therapy.
   2. Receipt of CAR-T-cell therapy or HCT either within 2 years of transplantation or receiving immunosuppressive therapy.
   3. Moderate or severe primary immunodeficiency (eg, DiGeorge syndrome, Wiskott-Aldrich syndrome).
   4. Use of at least 1 of the following immune-weakening medications:

      iii. Has received corticosteroids equivalent to prednisone ≥20 mg daily for at least 14 consecutive days within 30 days prior to study entry.

      iv. Active treatment causing significant immunosuppression, including alkylating agents, antimetabolites, transplant-related immunosuppressive drugs, cancer chemotherapeutic agents, TNF blockers, or other highly immunosuppressive drugs such as biologics.
   5. Hematological malignancy (including leukemia, lymphoma and myeloma) or active immunosuppressive treatment for solid tumor.
   6. HIV infection with CD4 cell count <200 mm3 from known medical history within the past 6 months of screening.
6. known severe renal impairment (eGFR of <30 mL/min/1.73 m2 within 6 months of the screening visit, using the serum creatinine-based CKD-EPI formula12).
7. Oxygen saturation of <92% on room air obtained at rest within 24h prior to randomization.
8. Has received or is expected to receive any other antiviral for the treatment of COVID 19, including remdesivir, PAXLOVID, molnupiravir, mAb treatment (within 30 days or 5 half-lives [whichever is longer] prior to screening) or received convalescent COVID-19 plasma within 12 months.
9. Expected to receive any dose of a SARS-CoV-2 vaccine within 14 days of randomization or during the study.
10. Current or previous administration with an investigational product (drug or vaccine) within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer). Authorized or products with conditional approval are not considered investigational.
11. Known prior participation in this trial
12. Known history of any of the following abnormalities in clinical laboratory tests (within past 6 months of the screening visit):

    * T bili ≥2 × ULN (except for Gilbert's syndrome)
    * AST or ALT ≥2.5 × ULN
    * Abs neutrophil count <1000/mm3.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (53):
- United States (53):
  - Cullman Clinical Trials, Cullman, Alabama
  - ClinMed, Phoenix, Arizona
  - Epic Medical Research - Surprise, Surprise, Arizona
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Franco Felizarta, Md, Bakersfield, California
  - Hope Clinical Research, Inc., Canoga Park, California
  - Velocity Clinical Research, Chula Vista, Chula Vista, California
  - Benchmark Research, Colton, California
  - Ascada Health PC dba Ascada Research, Fullerton, California
  - Long Beach Clinical Trials, Long Beach, California
  - Marvel Clinical Research - Santa Ana, Santa Ana, California
  - Herco Medical and Research Center Inc, Coral Gables, Florida
  - Advance Clinical Research Group, Cutler Bay, Florida
  - Proactive Clinical Research,LLC, Fort Lauderdale, Florida
  - Qway Research LLC, Hialeah, Florida
  - Unlimited Medical Research Group LLC, Hialeah Gardens, Florida
  - Angels Clinical Research Institute, Miami, Florida
  - South Florida Research Center, Miami, Florida
  - USPA Advance Concept Medical Research Group, Miami, Florida
  - Bio-Medical Research LLC, Miami, Florida
  - Coral Research Clinic Corp, Miami, Florida
  - Palm Springs Community Health Center, Miami Lakes, Florida
  - DBC Research USA, Pembroke Pines, Florida
  - GCP Research, Global Clinical professionals, St. Petersburg, Florida
  - Javara - Privia Medical Group Georgia - Albany, Albany, Georgia
  - Centricity Research Columbus Georgia Multispecialty, Columbus, Georgia
  - Centricity Research Columbus Acute Care, Columbus, Georgia
  - Rophe Adult and Pediatric Medicine/SKYCRNG, Union City, Georgia
  - Snake River Research, Idaho Falls, Idaho
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - Mercury Street Medical Group, PLLC, Butte, Montana
  - Henderson Clinical Trials, Henderson, Nevada
  - Excel Clinical Research, LLC, Las Vegas, Nevada
  - Monroe Biomedical Research, Monroe, North Carolina
  - Accellacare - Wilmington, Wilmington, North Carolina
  - Wellnow Urgent Care and Research, Cincinnati, Ohio
  - Remington-Davis, Inc, Columbus, Ohio
  - WellNow Urgent Care & Research, Dayton, Ohio
  - Kur Research @ Bon Secours Mercy Health, Inc - Urgent Care Easley, Easley, South Carolina
  - Javara - Privia Medical Group Gulf Coast - The Woodlands PGTW, Conroe, Texas
  - Javara - Privia Medical Group Gulf Coast - Cypress, Cypress, Texas
  - DFW Clinical Research, Dallas, Texas
  - Proactive Clinical Research LLC, Edinburg, Texas
  - Next Level Urgent Care, Houston, Texas
  - Laguna Clinical Research, Laredo, Texas
  - Epic Clinical Research, Lewisville, Texas
  - BFHC Research, LLC, San Antonio, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Javara - Privia Medical Group Gulf Coast - The Woodlands PGTW, Shenandoah, Texas
  - Javara - Privia Medical Group North Texas - Stephenville, Stephenville, Texas
  - Javara - Privia Medical Group Gulf Coast - The Woodlands PGTW, The Woodlands, Texas
  - Eastside Research Associates, Redmond, Washington

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Mortezavi M, Sloan A, Singh RSP, Chen LF, Kim JH, Shojaee N, Toussi SS, Prybylski J, Baniecki ML, Bergman A, Banerjee A, Allerton C, Alami NN. Virologic Response and Safety of Ibuzatrelvir, A Novel SARS-CoV-2 Antiviral, in Adults With COVID-19. Clin Infect Dis. 2025 Mar 17;80(3):673-680. doi: 10.1093/cid/ciae529. PMID 39486089
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5091003

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 278 participants were screened, of which 37 failed screening and 1 participant was not randomized due to investigational product shortage at site. A total of 240 participants were randomized and assigned to study intervention.
Groups:
- PF-07817883 100mg: Participants received PF-07817883, 100 milligrams (mg) orally every 12 hours (q12h) for 5 days (10 doses total). Participants were followed up for 4 weeks.
- PF-07817883 300mg: Participants received PF-07817883, 300 mg orally every q12h for 5 days (10 doses total). Participants were followed up for 4 weeks.
- PF-07817883 600mg: Participants received PF-07817883, 600 mg orally every q12h for 5 days (10 doses total). Participants were followed up for 4 weeks.
- Placebo: Participants received placebo orally every q12h for 5 days (10 doses total). Participants were followed up for 4 weeks.
Period: Treatment (Up to 5 Days)
Arm/Group | PF-07817883 100mg | PF-07817883 300mg | PF-07817883 600mg | Placebo
Started | 40 | 40 | 80 | 80
Treated | 40 | 39 | 79 | 79
Completed | 39 | 36 | 77 | 75
Not Completed | 1 | 4 | 3 | 5
Not completed — Adverse Event | 0 | 1 | 1 | 0
Not completed — Non-compliance with study drug | 0 | 0 | 0 | 1
Not completed — Other | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 3
Not completed — Randomized not treated | 0 | 1 | 1 | 1
Period: Follow Up (Up to 4 Weeks)
Arm/Group | PF-07817883 100mg | PF-07817883 300mg | PF-07817883 600mg | Placebo
Started | 39 | 37 (Eligible participants who discontinued study intervention could enter follow-up.) | 78 (Eligible participants who discontinued study intervention could enter follow-up.) | 76 (Eligible participants who discontinued study intervention could enter follow-up.)
Completed | 39 | 37 | 77 | 76
Not Completed | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention Participants were analyzed according to the intervention they were actually randomized.
Groups:
- PF-07817883 100mg: Participants received PF-07817883, 100 mg orally q12h for 5 days (10 doses total). Participants were followed up for 4 weeks.
- Total: Total of all reporting groups
Arm/Group | PF-07817883 100mg | PF-07817883 300mg | PF-07817883 600mg | Placebo | Total
Number analyzed (Participants) | 40 | 39 | 79 | 79 | 237
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.6 (12.30) | 41.9 (11.31) | 41.4 (11.60) | 41.5 (12.97) | 41.9 (12.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 29 | 50 | 45 | 147
  Male | 17 | 10 | 29 | 34 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 31 | 63 | 64 | 193
  Not Hispanic or Latino | 5 | 8 | 15 | 15 | 43
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 6 | 2 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 12 | 6 | 20
  White | 39 | 35 | 60 | 69 | 203
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Logarithm Base 10 (Log10) Transformed Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Ribo Nucleic Acid (RNA) Level on Day 5
Description: Change from baseline in SARS-CoV-2 RNA level at Day 5 was analyzed using Mixed Effects Repeated Measures (MMRM) model with fixed effects including treatment, visit, visit by treatment interaction, and baseline viral load. Covariates included days from baseline since symptom onset (<=3 versus [vs.] >3 days), vaccination status (complete or partial vs. unvaccinated), baseline anti-N serology status and age at screening (years). Participants were excluded from the analysis if baseline viral load was less than 4*log10 copies/milliliter, missing, or not detected.
Time Frame: Baseline (Day 1), Day 5
Population: The modified full analysis set (MFAS) included all participants in the full analysis set (FAS) who had SARS-CoV-2 RNA level greater than or equal to (>=) 4*log10 copies/mL at baseline. Participants were analyzed according to the study intervention to which they were randomized. Here 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (80% Confidence Interval); unit: Log10 copies/milliliter
Arm/Group | PF-07817883 100mg | PF-07817883 300mg | PF-07817883 600mg | Placebo
Number analyzed (Participants) | 34 | 24 | 66 | 60
Log10 copies/milliliter | -3.883 [-4.247 to -3.520] | -4.015 [-4.452 to -3.578] | -4.380 [-4.671 to -4.088] | -3.213 [-3.517 to -2.908]
Statistical Analysis 1: Comparison: PF-07817883 100mg vs Placebo; Test type: Other; p = 0.0181, Mixed Models Analysis; LS Mean difference = -0.671, 80% CI 2-sided [-1.080 to -0.262], Standard Error of Mean 0.3178
Statistical Analysis 2: Comparison: PF-07817883 300mg vs Placebo; Test type: Other; p = 0.0127, Mixed Models Analysis; LS Mean difference = -0.802, 80% CI 2-sided [-1.260 to -0.344], Standard Error of Mean 0.3562
Statistical Analysis 3: Comparison: PF-07817883 600mg vs Placebo; Test type: Other; p < .0001, Mixed Models Analysis; LS Mean difference = -1.167, 80% CI 2-sided [-1.506 to -0.827], Standard Error of Mean 0.2640

2. Secondary Outcome: Change From Baseline in Log10 Transformed SARS-CoV-2 RNA Level on Days 3, 10 and 14
Description: Change from baseline in SARS-CoV-2 RNA level at Day 3, Day 10 and Day 14 were analyzed using MMRM model with fixed effects including treatment, visit, visit by treatment interaction, and baseline viral load. Covariates included days from baseline since symptom onset (<=3 vs. >3 days), vaccination status (complete or partial vs. unvaccinated), baseline anti-N serology status and age at screening (years). Participants were excluded from the analysis if baseline viral load was less than 4*log10 copies/milliliter, missing, or not detected.
Time Frame: Baseline (Day 1), Day 3, Day 10 and Day 14
Population: The MFAS included all participants in the FAS who had SARS-CoV-2 RNA level >= 4*log10 copies/mL at baseline. Participants were analyzed according to the study intervention to which they were randomized. Here 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure. 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Least Squares Mean (80% Confidence Interval); unit: Log10 copies/milliliter
Arm/Group | PF-07817883 100mg | PF-07817883 300mg | PF-07817883 600mg | Placebo
Number analyzed (Participants) | 35 | 27 | 70 | 63
Log10 copies/milliliter
  Day 3 | -2.006 [-2.371 to -1.641] | -2.702 [-3.123 to -2.280] | -2.546 [-2.818 to -2.274] | -1.398 [-1.684 to -1.112]
  Day 10: number analyzed (Participants) | 32 | 27 | 68 | 57
  Day 10 | -5.027 [-5.326 to -4.728] | -5.085 [-5.423 to -4.748] | -5.305 [-5.529 to -5.082] | -5.091 [-5.332 to -4.851]
  Day 14: number analyzed (Participants) | 34 | 27 | 68 | 61
  Day 14 | -5.682 [-5.913 to -5.451] | -5.500 [-5.769 to -5.231] | -5.826 [-6.009 to -5.643] | -5.443 [-5.637 to -5.250]
Statistical Analysis 1: Comparison: PF-07817883 100mg vs Placebo; Day 3; Test type: Other; p = 0.0378, Mixed Models Analysis; LS Mean difference = -0.608, 80% CI 2-sided [-1.046 to -0.170], Standard Error of Mean 0.3402
Statistical Analysis 2: Comparison: PF-07817883 300mg vs Placebo; Day 3; Test type: Other; p = 0.0003, Mixed Models Analysis; LS Mean difference = -1.304, 80% CI 2-sided [-1.782 to -0.826], Standard Error of Mean 0.3718
Statistical Analysis 3: Comparison: PF-07817883 600mg vs Placebo; Day 3; Test type: Other; p < .0001, Mixed Models Analysis; LS Mean difference = -1.148, 80% CI 2-sided [-1.509 to -0.788], Standard Error of Mean 0.2803
Statistical Analysis 4: Comparison: PF-07817883 100mg vs Placebo; Day 10; Test type: Other; p = 0.5931, Mixed Models Analysis; LS Mean difference = 0.064, 80% CI 2-sided [-0.287 to 0.416], Standard Error of Mean 0.2732
Statistical Analysis 5: Comparison: PF-07817883 300mg vs Placebo; Day 10; Test type: Other; p = 0.5080, Mixed Models Analysis; LS Mean difference = 0.006, 80% CI 2-sided [-0.369 to 0.381], Standard Error of Mean 0.2914
Statistical Analysis 6: Comparison: PF-07817883 600mg vs Placebo; Day 10; Test type: Other; p = 0.1692, Mixed Models Analysis; LS Mean difference = -0.214, 80% CI 2-sided [-0.501 to 0.073], Standard Error of Mean 0.2230
Statistical Analysis 7: Comparison: PF-07817883 100mg vs Placebo; Day 14; Test type: Other; p = 0.1172, Mixed Models Analysis; LS Mean difference = -0.239, 80% CI 2-sided [-0.497 to 0.019], Standard Error of Mean 0.2004
Statistical Analysis 8: Comparison: PF-07817883 300mg vs Placebo; Day 14; Test type: Other; p = 0.3979, Mixed Models Analysis; LS Mean difference = -0.056, 80% CI 2-sided [-0.337 to 0.224], Standard Error of Mean 0.2178
Statistical Analysis 9: Comparison: PF-07817883 600mg vs Placebo; Day 14; Test type: Other; p = 0.0109, Mixed Models Analysis; LS Mean difference = -0.383, 80% CI 2-sided [-0.595 to -0.170], Standard Error of Mean 0.1655

3. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a study participant after administration of a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage. An adverse event is considered a treatment-emergent adverse event (TEAE) if the event started on or after the study medication start date and time. An SAE was any untoward medical occurrence at any dose that: resulted in death; was life-threatening (immediate risk of death); required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions) or resulted in congenital anomaly/birth defect or was considered an important medical event.
Time Frame: From start of study intervention up to 28 days after last dose of study intervention (up to 33 days)
Population: The safety analysis set (SAS) included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants were analyzed according to the intervention they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07817883 100mg | PF-07817883 300mg | PF-07817883 600mg | Placebo
Number analyzed (Participants) | 40 | 39 | 79 | 79
Participants
  TEAEs | 2 | 5 | 11 | 9
  SAEs | 0 | 1 | 0 | 0

4. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) Leading to Discontinuations
Description: An AE was any untoward medical occurrence in a study participant after administration of a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage. An adverse event is considered a treatment-emergent adverse event (TEAE) if the event started on or after the study medication start date and time. Participants with an AE record indicating the AE caused permanent discontinuation from the study were reported under discontinuations from study due to TEAEs. Permanent discontinuations from study intervention due to TEAEs included those participants who had an AE record that indicated that action taken with study treatment was drug withdrawn but AE did not cause the participant to be discontinued from study.
Time Frame: From start of study intervention up to 28 days after last dose of study intervention (up to 33 days)
Population: The SAS included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants were analyzed according to the intervention they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07817883 100mg | PF-07817883 300mg | PF-07817883 600mg | Placebo
Number analyzed (Participants) | 40 | 39 | 79 | 79
Participants
  Discontinuations from study due to TEAEs | 0 | 1 | 0 | 0
  Permanent discontinuations from study intervention due to TEAEs | 0 | 0 | 1 | 0

5. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: The following laboratory parameters were assessed according to pre-specified criteria for abnormalities: a) hematology; hemoglobin (gram per deciliter [g/dL]), (less than[<]0.8*lower limit of normal [LLN]), erythrocytes(10^12/Liter [L])(< 0.8*LLN), lymphocytes(10^9/L)(more than[>]1.2*upper limit of normal [ULN]), neutrophils(> 1.2*ULN and < 0.8*LLN), basophils(10^9/L)(> 1.2*ULN) and eosinophils (10^9/L)(> 1.2*ULN). b) clinical chemistry; bilirubin(mg/dL)(> 1.5*ULN), urea nitrogen(mg/dL)(> 1.3*ULN), creatinine(mg/dL)(> 1.3*ULN), potassium(milli equivalence per millilitre [mEq/L], (< 0.9*LLN and > 1.1*ULN), calcium (mg/dL)(< 0.9*LLN), bicarbonate(mEq/L)(< 0.9*LLN and > 1.1*ULN), glucose (mg/dL)(> 1.5*ULN), creatine kinase(units per litre [U/L) (> 2.0* ULN), D-Dimer(nanogram per milliliter[ng/mL]), (>1.5*ULN) and c)urinalysis; bacteria (low power field [LPF]>20). Number of participants with any laboratory abnormalities meeting pre-specified criteria are reported in this outcome measure.
Time Frame: From start of study intervention up to 28 days after last dose of study intervention (up to 33 days).
Population: The SAS included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants were analyzed according to the intervention they actually received. Here 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07817883 100mg | PF-07817883 300mg | PF-07817883 600mg | Placebo
Number analyzed (Participants) | 39 | 39 | 78 | 77
Participants | 4 | 4 | 18 | 13

6. Secondary Outcome: Number of Participants Meeting Pre-defined Criteria of Vital Sign Abnormalities
Description: Vital signs included blood pressure and pulse rate and were assessed with the participant in the supine or seated position with a completely automated device after at least 5 minutes of rest for the participant in a quiet setting without distractions. Pre-defined criteria for vital sign abnormalities was as systolic blood pressure (millimeter of mercury [mmHg]): value < 90, change >= 30 increase and change >= 30 decrease, diastolic blood pressure (mmHg): value <50; change >= 20 increase and change >= 20 decrease, pulse rate (beats per minute [bpm]): value < 40 and value > 120.
Time Frame: From start of study intervention up to 28 days after last dose of study intervention (up to 33 days).
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07817883 100mg | PF-07817883 300mg | PF-07817883 600mg | Placebo
Number analyzed (Participants) | 40 | 39 | 78 | 77
Participants
  Systolic blood pressure; value < 90 (mmHg) | 0 | 0 | 1 | 1
  Systolic blood pressure; change >= 30 (mmHg) increase | 0 | 0 | 1 | 0
  Systolic blood pressure; change >= 30 (mmHg) decrease | 1 | 2 | 0 | 3
  Diastolic blood pressure; value <50 (mmHg) | 0 | 0 | 0 | 0
  Diastolic blood pressure; change >= 20 (mmHg) increase | 1 | 1 | 1 | 2
  Diastolic blood pressure; change >= 20 (mmHg) decrease | 0 | 0 | 2 | 2
  Pulse rate; value < 40 (bpm) | 0 | 0 | 0 | 0
  Pulse rate; value > 120 (bpm) | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants Meeting Pre-defined Criteria For ECG Abnormalities
Description: Twelve lead ECGs were collected using an ECG machine that automatically calculated heart rate and measured PR interval, QT interval, and QT interval correct by Frederica formula (QTcF). ECG abnormalities included: PR interval (millisecond [msec]): value >=280, change >40 increase; QT interval aggregate (msec): value > 500), QTcF interval (450 < value =< 480; 480 < value =< 500; value > 500; 30 < change <= 60 increase and change > 60 increase).
Time Frame: From baseline (Day 1) up to Day 10
Population: The SAS included all participants randomly assigned to study intervention and who have taken at least 1 dose of study intervention. Participants were analyzed according to the intervention they actually received. Here 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07817883 100mg | PF-07817883 300mg | PF-07817883 600mg | Placebo
Number analyzed (Participants) | 40 | 39 | 79 | 78
Participants
  PR Interval, value >= 280 (msec) | 0 | 0 | 0 | 0
  PR Interval, change > 40 increase (msec) | 0 | 2 | 1 | 0
  QT Interval (msec) value >500 | 0 | 0 | 0 | 0
  QTcF Interval, 450 < value =< 480 (msec) | 1 | 1 | 2 | 6
  QTCF Interval, 480 < value =< 500 (msec) | 0 | 0 | 0 | 0
  QTCF Interval, value > 500 (msec) | 0 | 0 | 0 | 0
  QTCF Interval, 30 < change <= 60 increase (msec) | 5 | 6 | 6 | 9
  QTCF Interval, change > 60 increase (msec) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of study intervention up to 28 days after last dose of study intervention (up to 33 days).
Description: Same event may appear as both non-SAE and SAE but are distinct events. An event may be categorised as serious in 1 participant and non-serious in another, or a participant may have experienced both SAE and non-SAE.
Arm/Group | PF-07817883 100mg | PF-07817883 300mg | PF-07817883 600mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/39 | 0/79 | 0/79
Serious Adverse Events (participants affected / at risk) | 0/40 | 1/39 | 0/79 | 0/79
Other Adverse Events (participants affected / at risk) | 0/40 | 1/39 | 2/79 | 4/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-07817883 100mg (N=40) | PF-07817883 300mg (N=39) | PF-07817883 600mg (N=79) | Placebo (N=79)
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-07817883 100mg (N=40) | PF-07817883 300mg (N=39) | PF-07817883 600mg (N=79) | Placebo (N=79)
Alanine aminotransferase increased (Investigations) | 0 | 1 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-04-14): https://cdn.clinicaltrials.gov/large-docs/95/NCT05799495/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-12): https://cdn.clinicaltrials.gov/large-docs/95/NCT05799495/SAP_001.pdf